CLINICAL TRIAL: NCT04842201
Title: A Phase 1, Randomized, Placebo-Controlled, Double-blind, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of CM326 in Adult Healthy Volunteers
Brief Title: Single Ascending Dose Study of CM326 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CM326HV001
Record Dates: First submitted 2021-04-08; First posted 2021-04-13 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2021-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CM326 (Experimental): subcutaneous injection
  Interventions: Drug: CM326
- Placebo (Placebo Comparator): subcutaneous injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CM326 — subcutaneous injection
  Arms: CM326
Drug: Placebo — subcutaneous injection
  Arms: Placebo

SUMMARY:
Single ascending dose study to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics and immunogenicity of CM326 in healthy volunteers.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy adult male participant,18 to 65 years of age, inclusive.
* Body Mass Index (BMI) 18 to 26 kg/m2, inclusive.
* History, physical examination, laboratory tests and test related items of inspection were normal or abnormal without clinically insignificant.
* Males must abstain from sex or use highly effective methods of birth control.
* Having given written informed consent prior to undertaking any study-related procedure.

Key Exclusion Criteria:

* Positive for HIV, or Hepatitis B, or C.
* Positive result on urine drug screen.
* Clinical laboratory abnormalities of clinical significance, or other clinical findings suggest clinically significant following diseases (including, but not limited to the gastrointestinal tract, kidney, liver, nerve, blood, endocrine, cancer, lung, immune, mental or cardiovascular disease).
* With any condition that inappropriate for entry into this study.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2021-09-28 (Actual); Study Completion 2021-09-28 (Actual)

PRIMARY OUTCOMES:
Safety of CM326 by assessing the number and severity of adverse events, including changes in vital signs, physical examination, laboratory safety tests, and ECGs | Day 1 through Day 85

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of CM326 | Day 1 through Day 85
  Serum concentrations of CM326 over time
Pharmacodynamics of CM326 | Day 1 through Day 85
  Serum total Immunoglobulin E (IgE) and Thymus and activation regulated chemokine (TARC) over time
Immunogenicity | Day 1 through Day 85
  anti-drug antibody (ADA)

CONTACTS AND LOCATIONS:
Overall Officials: Jie Hou, Principal Investigator — Peking University Care Luzhong Hospital
Locations (1):
- PKUCare Luzhong Hospital, Zibo, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Di Y, Yang L, Zhou J, Zhang L, Huang Y, Jia Y, Yan H, Chen L, Hou Q, Chen B, Luo Z, Hou J. Translational Investigation of CM326 from Preclinical Studies to Randomized Phase I Clinical Trials in Healthy Adults. BioDrugs. 2025 May;39(3):487-498. doi: 10.1007/s40259-025-00714-4. Epub 2025 Apr 4. PMID 40185989